CLINICAL TRIAL: NCT03989011
Title: Tonometry (1) and Duplex Ultrasound (2) to Predict Abdominal Aorta Aneurysm (3) Progression and Cardiovascular Events in Aneurysm Patients
Brief Title: Tonometry and Duplex Ultrasound to Predict AAA Progression and CV Events in Aneurysm Patients (1-2-3 Trial)
Status: Completed | Type: Observational
Sponsor: Rijnstate Hospital (Other)
Collaborators: Radboud University Medical Center (Other); Canisius-Wilhelmina Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: NL68953.091.19
Record Dates: First submitted 2019-05-29; First posted 2019-06-18 (Actual); Last update posted 2024-04-11 (Actual); Status verified 2024-04

CONDITIONS: Abdominal Aortic Aneurysm; Cardiovascular Events
Keywords: Functional response; Abdominal Aortic Aneurysm; Cardiovascular events
MeSH Terms: conditions — Aortic Aneurysm, Abdominal | interventions — Vascular Stiffness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Carotid Artery Reactivity test (CAR test) — The CAR test will be applied to stimulate the sympathetic nervous system. This thermal stimulus is known to elevate blood pressure via sympathetic pathways, so it can be used to study the vascular response to sympathetic activation. The participant will submerge their left hand in a bucket of ice water (approximately 4 degrees celsius) for 3 minutes, which is reported to be sufficient to induce a maximal dilation in the common carotid artery. At baseline and every minute after the hand is submerged in ice water, the blood pressure will be measured to check whether a sympathetic stimulation is achieved.
Diagnostic Test: Arterial stiffness — The SphygmoCor device will be used to non-invasively measure arterial stiffness parameters using applanation tonometry. For Pulse Wave Analyses (PWA), the radial waveform will be recorded. Approximately 10 waveforms are averaged, resulting in several non-invasive parameters:
  * Peripheral pressure parameters
  * Central and abdominal aneurysm pressure parameters (derived using a transfer function)
  * Cardiac output parameters (SEVR, ED)
  Pulse wave velocity will be performed by recording the waveforms of the carotid and femoral artery sequentially. The travelled distance will be measured according to the current guidelines and entered in the program. The program will calculate the PWV based on 10 ECG triggered waveform of each artery.

SUMMARY:
Abdominal aortic aneurysm (AAA) is a common vascular disease and associated with risk of rupture, but also with a high cardiovascular (CV) event rate. A key difficulty in AAA is predicting these life-threatening complications, highlighting the need to explore the potential of novel techniques. Both progression of AAA and CV events are strongly linked to vascular health. In 2013, the SMART risk score is developed to calculate the risk of the patients for recurrent vascular events based on clinical characteristics. Recently, a novel, easy to perform, non-invasive test of endothelial function (the carotid artery reactivity (CAR) test), reflecting target organ damage, has recently been introduced. The CAR is a simple, quick (5-min), non-invasive test that uses ultrasound to examine the carotid artery in response to sympathetic stimulation by placing one hand in cold water. This test shows strong agreement with both coronary and aortic responses to sympathetic stimulation and predicted CV events in patients with peripheral arterial disease.

The aim of this prospective 2-year follow-up study is to investigate the predictive capacity of the CAR-test in comparison to the SMART risk score for the development of cardiovascular events in patients with an abdominal aortic aneurysm who have not yet reached the treatment threshold. This could aid clinical decision making in the need for (surgical) intervention, but also alter (drug) treatment to reduce risk of cardiovascular events. Secondary objectives are to investigate the predictive capacity of the CAR-test for progression of the abdominal aortic aneurysm, and to evaluate QoL scores in patients under surveillance for AAA. The aim is to provide insight if these scores can help clinical decision making.

DETAILED DESCRIPTION:
The investigators will include 167 patients under surveillance for AAA who are all currently under the threshold for repair (i.e. AAA diameter 40-50 mm for men and 35-45 mm for women). Participants will be recruited from all collaborating hospitals (Radboudumc, Rijnstate, CWZ) after providing written informed consent. Additionally, AAA-patients under surveillance of general practitioners are eligible (and will be contacted through the hospital-links), since the nature of the tests allow for performing all tests at the general practitioners' office.

In this observational, prospective study, a total of 167 patients under surveillance for an AAA, who are currently under threshold for repair (i.e. AAA diameter 40-50 mm for men and 35-44 mm for women), will be included. Baseline patient characteristics will be registered, including traditional risk factors and CV-history. In addition to regular care of measuring AAA diameter progression (in mm/year), the investigators will perform the CAR-test (10-min) and non-invasive arterial stiffness measures (PWA and PWV with the SphygmoCor device (10-min) one time as baseline. Furthermore, the investigators will ask patients to complete a questionnaire about the quality of their life (Appendix 1). A second questionnaire tries to clarify the disease experience of the patients and can be found in Appendix 2. Both questionnaires will be asked to be completed at the start and the end of the study. Subsequently, the investigators will record major adverse cardiovascular events (MACE) according to the International Classification of Disease-10. Registration of MACE will be performed using hospital-records and following international guidelines. Across a 2-year follow-up, by means of regular follow-up appointments, the investigators will examine AAA progression (in mm/year) and the ability of the CAR parameter and arterial stiffness parameters to predict CV-events.

ELIGIBILITY:
Inclusion Criteria:

* Male or female at least 18 years old;
* Informed consent form understood and signed and patient agrees to follow- up visits;
* Has an abdominal aortic aneurysm (AAA), who is still under surveillance;

Exclusion Criteria:

* Life expectancy < 2 years;
* Psychiatric or other condition that may interfere with the study;
* Participating in another clinical study, interfering on outcomes;
* Increased risk for coronary spasms (score Rose-questionnaire ≥2; this questionnaire can be found in Appendix 3);
* Presence of Raynaud's phenomenon, chronic pain syndrome at upper extremity(s), presence of an AV fistula or shunt, open wounds to the upper extremity(s), and/or scleroderma associated with placing the hand in ice water;
* Recent (<3 months) presence of angina pectoris, myocardial infarction, cerebral infarction, and/or heart failure, or PAD treatment.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients under surveillance for an AAA, who are currently under threshold for repair (i.e. AAA diameter 40-50 mm men and 35-44 mm for women), will be included. AAA patients will be recruited from all collaborating hospitals (Radboudumc, Rijnstate, CWZ), who provide written informed consent. Additionally, also AAA-patients under surveillance of general practitioners are eligible (and will be contacted through the hospital-links), since the nature of the tests allow for performing all tests at the general practitioners' office.
Sampling Method: Non-Probability Sample
Enrollment: 167 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2023-05-01 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
Major Adverse Cardiovascular Events (MACE) | 2 year follow-up
  Incidence of MACE including myocardial infarction, cerebral infarction, heart failure, and peripheral vascular disease

SECONDARY OUTCOMES:
SMART risk score | Baseline
  Second Manifestations of ARTerial disease risk score is developed to determine the risk of recurrent vascular events based on clinical characteristics of the patients
SphygmoCor parameters | Baseline
  Peripheral pressure measurements (PWA)
SphygmoCor parameters | Baseline
  central pressure measurements (derived using a transfer function, PWA)
SphygmoCor parameters | Baseline
  abdominal pressure measurements (derived using a transfer function, PWA)
SphygmoCor parameters - cardiac output parameter | Baseline
  SEVR
SphygmoCor parameters - cardiac output parameter | Baseline
  ED
SphygmoCor parameters | Baseline
  PWV
CAR-test results | Baseline
  Percentage of vasodilation/vasoconstriction to the CAR test at the common carotid artery at baseline
CAR-test results | Baseline
  magnitude of the blood flow and perfusion response
CAR-test results | Baseline
  timing of the blood flow and perfusion response
CAR-test results | Baseline
  blood pressure responses
CAR-test results | Baseline
  heart rate responses
AAA progression | 2 year follow up
  AAA diameter progression in mm/year
Aorta repair | Within 2 year follow-up
  If the patient underwent aorta repair
AAA rupture | Within 2 year follow up
  If the AAA ruptured
Score EQ-5D questionnaire | At baseline and after 2 years
  Patient reported outcomes measured by the general health questionnaire
Score IPQ-K questionnaire | At baseline and after 2 years
  Patient reported outcomes measured by the disease perception questionnaire
Clinical success | 2 year follow up
  Incidence of serious adverse events

OTHER OUTCOMES:
Demographic characteristics | 2 year follow up
  Age
Demographic characteristics | 2 year follow up
  gender
Demographic characteristics | 2 year follow up
  height
Demographic characteristics | 2 year follow up
  weight
Demographic characteristics | 2 year follow up
  ASA class
Demographic characteristics | 2 year follow up
  medical history
Demographic characteristics | 2 year follow up
  blood pressure
Demographic characteristics | 2 year follow up
  heart rate
Demographic characteristics | 2 year follow up
  cardiac measurements
Demographic characteristics | 2 year follow up
  SVS class
Medication use | 2 year follow up
  Anti-platelets
Medication use | 2 year follow up
  anti-coagulants
Medication use | 2 year follow up
  anti-hypertensives
Medication use | 2 year follow up
  statins
Medication use | 2 year follow up
  beta-blockers
Medication use | 2 year follow up
  sympathicomimetics
Laboratory results | 2 year follow up
  Hemoglobin
Laboratory results | 2 year follow up
  serum creatinine
Laboratory results | 2 year follow up
  cholesterol
Laboratory results | 2 year follow up
  eGFR
Laboratory results | 2 year follow up
  crp
Anatomic characteristics of AAA | 2 year follow up
  AAA sac diameter
Anatomic characteristics of AAA | 2 year follow up
  infrarenal aortic neck lumen diameter
Anatomic characteristics of AAA | 2 year follow up
  proximal non-aneurysmal aortic neck length
Anatomic characteristics of AAA | 2 year follow up
  proximal aortic neck angle
Anatomic characteristics of AAA | 2 year follow up
  aneurysm blood lumen diameter
Anatomic characteristics of AAA | 2 year follow up
  common iliac artery diameter left
Anatomic characteristics of AAA | 2 year follow up
  common iliac artery diameter right
Anatomic characteristics of AAA | 2 year follow up
  blood lumen diameter

CONTACTS AND LOCATIONS:
Overall Officials: Michel Rijnen, MD, prof, Principal Investigator — Rijnstate Hospital
Locations (3):
- Netherlands (3):
  - Radboudumc, Nijmegen, Gelderland
  - Canisius Wilhelmina Ziekenhuis, Nijmegen, Gelderland
  - Rijnstate Hospital, Arnhem